CLINICAL TRIAL: NCT02677740
Title: Mechanisms of Non-Invasive Neuromodulation Interventions: Influence on Human Neurochemistry and Functional Connectivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1601M83405
Record Dates: First submitted 2016-02-02; First posted 2016-02-09 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Non-invasive Neuromodulation in Healthy Subjects
Keywords: MRI; MRS; rTMS

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Inhibitory rTMS (1 Hz) (Experimental): Subjects are exposed to a 20-min inhibitory rTMS intervention that transiently suppresses the excitability of cortical structures beneath the site of stimulation. Subjects undergo MRI and MRS both before and right after the rTMS intervention.
  Interventions: Device: Inhibitory rTMS (1 Hz)
- Excitatory rTMS (5 Hz) (Experimental): Subjects are exposed to a 20-min excitatory rTMS intervention that transiently increases the net excitability of cortical structures beneath the site of stimulation. Subjects undergo MRI and MRS both before and right after the rTMS intervention.
  Interventions: Device: Excitatory rTMS (5 Hz)

INTERVENTIONS:
Device: Inhibitory rTMS (1 Hz) — Participants receive rTMS at a rate of 1 Hz, applied with a 70-mm figure-eight TMS coil connected to a stimulator, over the motor cortex hotspot contralateral to the dominant arm for 20 minutes at an intensity of 90% resting motor threshold (RMT) for a total of 600 TMS pulses. The total number of stimuli applied is well within the published safety guidelines for use of rTMS. rTMS is applied outside the scanner, whereas functional connectivity and neurochemistry are measured with MRI and MRS, respectively, at 7 Tesla. The MRI/MRS data are collected right before and immediately after the inhibitory rTMS intervention.
  Arms: Inhibitory rTMS (1 Hz)
Device: Excitatory rTMS (5 Hz) — Participants receive rTMS at a rate of 5 Hz, applied with a 70-mm figure-eight TMS coil connected to a stimulator, over the motor cortex hotspot contralateral to the dominant arm for 20 minutes at an intensity of 90% RMT for a total of 600 TMS pulses. The total number of stimuli applied is well within the published safety guidelines for use of rTMS. rTMS is applied outside the scanner, whereas functional connectivity and neurochemistry are measured with MRI and MRS, respectively, at 7 Tesla. The MRI/MRS data are collected right before and immediately after the excitatory rTMS intervention.
  Arms: Excitatory rTMS (5 Hz)

SUMMARY:
The aim of this project is to increase our understanding of how two different protocols of repetitive transcranial magnetic stimulation (rTMS), inhibitory (1 Hz) and excitatory (5 Hz), applied over the primary motor cortex of the presumed dominant hemisphere, affect functional connectivity and neurochemistry in the brain.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation method which is effective for treating both psychiatric and non-psychiatric disorders, such as posttraumatic stress disorder, obsessive compulsive disorder, pain syndromes and for improving motor function in neurodegenerative diseases or following stroke. rTMS uses series of brief pulses of magnetic field applied to the surface of the head for a period of time (e.g. 20 minutes). The effects of rTMS are transient, and critically dependent upon the location, frequency and intensity of stimulation. Several studies have provided evidence that rTMS can influence the excitability and function of neurons (neuromodulation) for up to one hour, both near to, and distant from, the site of stimulation. However it is still unclear how these transient local and distant changes in function induced by specific rTMS protocols are mediated. In this project we will combine expertise in Magnetic Resonance Imaging (MRI), Magnetic Resonance Spectroscopy (MRS) and rTMS neuromodulation to develop and test protocols for examining the changes produced by non-invasive brain stimulation on healthy subjects. rTMS will be applied outside the scanner using standard TMS coils and MRI/S at 7 Tesla will be acquired before and immediately after rTMS. Our aim is to increase the understanding of how the two different rTMS protocols, inhibitory (1 Hz) and excitatory (5 Hz), applied over the primary motor cortex of the presumed dominant hemisphere, affect functional connectivity and neurochemistry in the brain.

ELIGIBILITY:
Inclusion Criteria:

Those volunteers who are evaluated as normal and not met exclusion criteria will be potential candidates for this study.

Exclusion Criteria:

The following participants will be excluded from this study, including but not limited to:

* Females
* Left handed males
* Participants who never underwent MRI at 7 Tesla

Participants with:

* any type of bio-implant activated by mechanical, electronic, or magnetic means (e.g. cochlear implants, pacemakers, neurostimulators, bio stimulators, electronic infusion pumps.)
* any type of ferromagnetic bio-implant that could potentially be displaced or damaged, such as aneurysm clips, metallic skull plates, etc.
* non-removable piercing or permanent eyeliner
* retained metal in their body, either from a medical procedure or an injury

Participants who:

* have been diagnosed by a physician as having a psychiatric disorder, substance abuse, neurological and/or cardiovascular disease
* have cardiac or known circulatory impairment, and/or the inability to perspire (poor thermoregulatory function)
* have hyper- or hypotension or arrhythmias
* have known conditions which can lead to emergency medical care
* had a head injury that caused them to lose consciousness for more than 30 minutes or have amnesia for more than 24 hours
* had a brain tumor or stroke
* had one or more seizures, or been given a diagnosis of epilepsy
* have a history of sleep apnea or head trauma that may have caused Traumatic Brain Injury (TBI)
* have a history of anxiety, syncope, panic attacks and/or claustrophobia
* cannot adhere to the experimental protocol for any reason
* started taking chemotherapy or immunomodulatory agents, or had any radiation treatment that could affect the brain
* are currently on any medication

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2017-03-19 (Actual); Study Completion 2017-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Mangia, PhD, Principal Investigator — Dept. of Radiology, University of Minnesota
Locations (1):
- Center for Magnetic Resonance Research, Dept. of Radiology, University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Emara TH, Moustafa RR, ElNahas NM, ElGanzoury AM, Abdo TA, Mohamed SA, ElEtribi MA. Repetitive transcranial magnetic stimulation at 1Hz and 5Hz produces sustained improvement in motor function and disability after ischaemic stroke. Eur J Neurol. 2010 Sep;17(9):1203-1209. doi: 10.1111/j.1468-1331.2010.03000.x. Epub 2010 Apr 8. PMID 20402755
- [Background] Machado S, Bittencourt J, Minc D, Portella CE, Velasques B, Cunha M, Budde H, Basile LF, Chadi G, Cagy M, Piedade R, Riberio P. Therapeutic applications of repetitive transcranial magnetic stimulation in clinical neurorehabilitation. Funct Neurol. 2008 Jul-Sep;23(3):113-22. PMID 19152730
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Bednarik P, Tkac I, Giove F, DiNuzzo M, Deelchand DK, Emir UE, Eberly LE, Mangia S. Neurochemical and BOLD responses during neuronal activation measured in the human visual cortex at 7 Tesla. J Cereb Blood Flow Metab. 2015 Mar 31;35(4):601-10. doi: 10.1038/jcbfm.2014.233. PMID 25564236
- [Background] Smith SM, Beckmann CF, Andersson J, Auerbach EJ, Bijsterbosch J, Douaud G, Duff E, Feinberg DA, Griffanti L, Harms MP, Kelly M, Laumann T, Miller KL, Moeller S, Petersen S, Power J, Salimi-Khorshidi G, Snyder AZ, Vu AT, Woolrich MW, Xu J, Yacoub E, Ugurbil K, Van Essen DC, Glasser MF; WU-Minn HCP Consortium. Resting-state fMRI in the Human Connectome Project. Neuroimage. 2013 Oct 15;80:144-68. doi: 10.1016/j.neuroimage.2013.05.039. Epub 2013 May 20. PMID 23702415
- See also: Profile of Principal Investigator — http://www.cmrr.umn.edu/facultystaff/mangia.shtml

RESULTS

PARTICIPANT FLOW:
Groups:
- Inhibitory rTMS (1 Hz): Subjects are exposed to a 20-min inhibitory rTMS intervention that transiently suppresses the excitability of cortical structures beneath the site of stimulation. Subjects undergo MRI and MRS both before and right after the rTMS intervention. One week before the MRI/MRS acquisitions, neurophysiological parameters are also measured before and right after the rTMS intervention.
  Inhibitory rTMS (1 Hz): Participants receive rTMS at a rate of 1 Hz, applied with a 70-mm figure-eight TMS coil connected to a stimulator, over the motor cortex hotspot contralateral to the dominant arm for 20 minutes at an intensity of 90% resting motor threshold (RMT) for a total of 600 TMS pulses. The total number of stimuli applied is well within the published safety guidelines for use of rTMS. rTMS is applied outside the scanner, whereas functional connectivity and neurochemistry are measured with MRI and MRS, respectively, at 7 Tesla. The MRI/MRS data are collected right before and immediately after the
- Excitatory rTMS (5 Hz): Subjects are exposed to a 20-min excitatory rTMS intervention that transiently increases the net excitability of cortical structures beneath the site of stimulation. Subjects undergo MRI and MRS both before and right after the rTMS intervention. One week before the MRI/MRS acquisitions, neurophysiological parameters are also measured before and right after the rTMS intervention.
  Excitatory rTMS (5 Hz): Participants receive rTMS at a rate of 5 Hz, applied with a 70-mm figure-eight TMS coil connected to a stimulator, over the motor cortex hotspot contralateral to the dominant arm for 20 minutes at an intensity of 90% RMT for a total of 600 TMS pulses. The total number of stimuli applied is well within the published safety guidelines for use of rTMS. rTMS is applied outside the scanner, whereas functional connectivity and neurochemistry are measured with MRI and MRS, respectively, at 7 Tesla. The MRI/MRS data are collected right before and immediately after the excitatory rTMS interv
Period: Overall Study
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz)
Started | 7 | 1
Completed | 7 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz) | Total
Number analyzed (Participants) | 7 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 1 | 8
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (7) | 22 (NA) — There is only one participant in this arm, therefore, the standard deviation cannot be calculated. | 27 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 1 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 1 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percent Change of GABA Concentration in a Voxel Encompassing the Left Motor Cortex, Measured at 30 Min After rTMS
Description: GABA concentration is quantified with MRS at 7 Tesla. Percent change of GABA concentration is calculated from baseline (i.e., pre-rTMS).
Time Frame: Baseline/Pre-rTMS and 30 min after rTMS
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz)
Number analyzed (Participants) | 7 | 1
percent change | 8 (9) | -27 (NA) — There is only one participant in this arm, therefore, the standard deviation cannot be calculated.

2. Primary Outcome: Percent Change of GABA Concentration in a Voxel Encompassing the Right Motor Cortex, Measured at 60 Min After rTMS
Description: as for outcome 1
Time Frame: Baseline/Pre-rTMS and 60 min after rTMS
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz)
Number analyzed (Participants) | 7 | 1
percent change | -6 (6) | 4 (NA) — There is only one participant in this arm, therefore, the standard deviation cannot be calculated.

3. Primary Outcome: Percent Change of Functional Connectivity in Left Motor Cortex, Where Functional Connectivity is Measured as a Dimensionless Fractional Amplitude of Low-frequency Fluctuations (fALFF), at 80 Min After rTMS
Description: Functional connectivity is measured with MRI at 7 Tesla as a dimensionless fractional amplitude of low-frequency fluctuations (fALFF). This is an index which reflects the intensity of spontaneous regional brain activity. It is calculated as the ratio of power spectra of low frequency (0.01-0.08 Hz) to that of the entire frequency range. Percent change of functional connectivity is calculated from baseline (i.e., pre-rTMS).
Time Frame: Baseline/Pre-rTMS and 80 min after rTMS
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz)
Number analyzed (Participants) | 7 | 1
percent change | -2 (11) | 9 (NA) — There is only one participant in this arm, therefore, the standard deviation cannot be calculated.

4. Primary Outcome: Percent Change of Functional Connectivity in Right Motor Cortex, Where Functional Connectivity is Measured as a Dimensionless Fractional Amplitude of Low-frequency Fluctuations (fALFF), at 80 Min After rTMS
Description: as for outcome 3
Time Frame: Baseline/Pre-rTMS and 80 min after rTMS
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz)
Number analyzed (Participants) | 7 | 1
percent change | -1 (10) | 17 (NA) — There is only one participant in this arm, therefore, the standard deviation cannot be calculated.

ADVERSE EVENTS:
Time Frame: approximately 4 hours
Arm/Group | Inhibitory rTMS (1 Hz) | Excitatory rTMS (5 Hz)
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/1
Other Adverse Events (participants affected / at risk) | 7/7 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inhibitory rTMS (1 Hz) (N=7) | Excitatory rTMS (5 Hz) (N=1)
Sleepiness (General disorders) | 3 (3) | 1 (1)
Warmth (General disorders) | 1 (1) | 0 (0)
Metallic Taste (General disorders) | 1 (1) | 1 (1)
Anxiety/Worry/Nervousness (Psychiatric disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 1 (1) | 0 (0)
Tooth Pain (General disorders) | 1 (1) | 0 (0)
Shoulder Pain (General disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was initially registered with a larger number of subjects (30) than what the pilot funds allowed (8) to allow more studies in the future. However, we decided to close the protocol after 8 studies reported here to avoid prolonged inactivity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT02677740/Prot_SAP_000.pdf